CLINICAL TRIAL: NCT02937519
Title: Multi-center Phase II Clinical Randomized Study of Chronomodulated Chemotherapy Followed by Concurrent Chemo-radiotherapy With IMRT in the Treatment of Advanced Nasopharyngeal Cancer
Brief Title: Chronomodulated Chemotherapy Followed by Concurrent Chemo-radiotherapy With IMRT in the Treatment of Advanced Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyang Medical University (Other)
Collaborators: The Affiliated Cancer Hospital of Xiangya School of Medicine Central South University (Unknown); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Feng Jing, Chief physician/Professor, Guiyang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016080201
Record Dates: First submitted 2016-08-16; First posted 2016-10-18 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Esophageal Neoplasms
Keywords: Chronomodulated Chemotherapy; Intensity Modulated Radiation Therapy; Advanced Nasopharyngeal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melodie group (Experimental): Induction chrono-chemotherapy followed by cisplatin chrono-chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Device: Chrono-chemotherapy pump:Melodie; Drug: induction Chrono-chemotherapy; Drug: cisplatin chrono-chemotherapy; Radiation: intensity-modulated radiation therapy
- Routine-Chemotherapy (Other): Induction routine-chemotherapy followed by cisplatin routine-chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Device: Routine intravenous drip; Drug: induction Routine-chemotherapy; Drug: cisplatin routine-chemotherapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Device: Chrono-chemotherapy pump:Melodie
  Arms: Melodie group
Device: Routine intravenous drip
  Arms: Routine-Chemotherapy
Drug: induction Chrono-chemotherapy
  Arms: Melodie group
Drug: induction Routine-chemotherapy
  Arms: Routine-Chemotherapy
Drug: cisplatin chrono-chemotherapy
  Arms: Melodie group
Drug: cisplatin routine-chemotherapy
  Arms: Routine-Chemotherapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
1. Observe and compare the chrono-chemotherapy IMRT and conventional chemotherapy and intensity modulated radiotherapy term efficacy of the treatment of locally advanced nasopharyngeal carcinoma.
2. Evaluation chrono-chemotherapy IMRT and conventional chemotherapy and intensity modulated radiotherapy in locally advanced nasopharyngeal carcinoma safety and tolerability.

3）observing the adverse reaction and effects of two groups,expected chrono-chemotherapy group can achieve lower toxicity, improve the curative effect, for the treatment of nasopharyngeal carcinoma provides a more reasonable way.

ELIGIBILITY:
Inclusion Criteria:

* initial treatment of advanced nasopharyngeal carcinoma Ⅲ-Ⅳ patients with pathologically confirmed (according to 2010 UICC staging, T3-4, N0-3), without evidence of distant metastasis (M0). Have measurable tumor lesions.
* KPS≥70 points.
* the age of 18-70 years old, male or female.
* no major organ dysfunction; normal bone marrow function (WBC ≥4.0 × 109 / L, platelets ≥100 × 109 / L, hemoglobin ≥90g / L), normal liver function (total bilirubin, alanine aminotransferase, aspartate aminotransferase ≤1.5 times the upper limit of normal), normal renal function (creatinine ≤ 1.5 times upper limit of normal).
* understand this study and signed informed consent.

Exclusion Criteria:

* distant metastasis.
* who had received prior chemotherapy.
* patients have physical or mental illness, and by researchers believe that patients can not be completely or fully understood in this study possible complications.
* pregnancy (via the urine or serum β-HCG test confirmed) or during lactation.
* serious complications, such as uncontrolled hypertension, heart failure, diabetes and so on.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with curative effect | 1 year
  Evaluate the immediate effect at 1year after Concurrent chemo-radiotherapy by RECIST.
Number of Participants with Adverse Events as a Measure of Safety | 5 years
  To assess and record nausea, vomiting, oral mucositis, diarrhea and other adverse drug reactions by CTC 3.0.

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Evaluate the Progression-free survival at five years after Concurrent chemo-radiotherapy by RECIST.
Overall survival | 5 years
  Evaluate the Overall survival at five years after Concurrent chemo-radiotherapy by RECIST.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes